CLINICAL TRIAL: NCT06405217
Title: Safety and Efficacy of Recombinant Human Thyroid Stimulating Hormone for Radioiodine 131I Treatment in Patients With Locally Advanced/Metastatic Differentiated Thyroid Cancer
Brief Title: Recombinant Human Thyroid Stimulating Hormone for Radioiodine 131I Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Feng Wang, Director of nuclear medicine department, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20240419-09
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: DTC - Differentiated Thyroid Cancer; Thyroid Stimulating; Hormone, C; Radiotherapy; Complications
MeSH Terms: interventions — Thyrotropin Alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant human thyroid stimulating hormone group (Experimental): Recombinant human thyroid stimulating hormone injection: 0.9mg/1.0mL/piece; intramuscular injection; once a day for two consecutive days
  Interventions: Drug: Recombinant Human Thyroid Stimulating Hormone
- Withdraw group (No Intervention): Thyroid hormone withdraw for 4-6 weeks

INTERVENTIONS:
Drug: Recombinant Human Thyroid Stimulating Hormone — Recombinant human thyroid stimulating hormone injection: 0.9mg/1.0mL/piece; intramuscular injection; once a day for two consecutive days
  Arms: Recombinant human thyroid stimulating hormone group

SUMMARY:
Subjects: patients with postoperative local recurrent or metastatic differentiated thyroid cancer .

Experimental group: Recombinant human thyroid stimulating hormone injection: 0.9mg/1.0mL/piece; intramuscular injection; once a day for two consecutive days. Control group: Thyroid hormone withdraw for 4-6 weeks.

The two groups were treated with radioiodine 131I after plasma thyroid stimulating hormone elevated (>30mU/L). The efficacy and adverse reactions were observed.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18~75 years old (including 18 and 75 years old);
* ECOG: 0-2 points;
* Expected survival of more than 3 months; Differentiated thyroid carcinoma undergoing total thyroidectomy or subtotal thyroidectomy and confirmed as locally recurrent or metastatic disease by imaging, serum tumor marker, biopsy pathology; at least one measurable lesion (diameter of the tumor ≥10 mm), and meets the requirements of RECIST 1.1.
* Hemoglobin ≥80g/L, neutrophil ≥1.5×109/L, platelet count ≥80×109/L, serum creatinine ≤1.5× upper limit of normal or creatinine clearance ≥60ml/min, Blood urea nitrogen ≤2.5× upper limit of normal (ULN); Total bilirubin ≤1.5×ULN; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN; If accompanied by liver metastasis, ALT and AST≤5×ULN albumin ≥25 g/L;
* Women of childbearing potential must have taken reliable contraceptive measures or undergone a pregnancy test (serum or urine) within 7 days prior to enrollment, with a negative result, and be willing to use appropriate contraceptive methods during the trial and for 1 year after the last dose of 131I (for women), or for 6 months after the last dose of 131I (for men);
* Participants voluntarily joined the study and signed informed consent, with good compliance and follow-up.

Exclusion Criteria:

* Patients with severe and uncontrolled diseases, including: 1) Uncontrolled hypertension (despite optimal drug therapy, systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg); 2) Poorly controlled arrhythmias of ischemic heart disease or myocardial infarction of grade II or above (including corrected QT interval male ≥450 ms, female ≥470 ms) and ≥2 congestive heart failures (New York Heart Association classification); 3) Poorly controlled diabetes (fasting blood sugar >10mmol/L); 4) Active or poorly controlled severe infections (according to Common Terminology Criteria for Adverse Events ≥ grade 2); 5) Patients with active hepatitis B or hepatitis C (hepatitis B: positive HBsAg and hepatitis B virus (HBV) DNA ≥500 IU/mL; hepatitis C: positive hepatitis C virus RNA and abnormal liver function), or active infections requiring antimicrobial therapy (e.g., with antibiotics, antiviral drugs, antifungal drugs); 6) Renal insufficiency: urine routine shows urine protein ≥++ or confirmed 24-hour urine protein ≥1.0 g; 7) Patients with seizures requiring treatment.
* Received surgical treatment, incisional biopsy, or major trauma within 28 days prior to randomization;
* Unable to quit or with a history of psychiatric medication abuse;
* Allergic to the investigational drug (recombinant human thyroid stimulating hormone or 131I) or its excipients;
* Had an infection within 4 weeks prior to screening, including bacterial, viral, or fungal infections, with ongoing symptoms at the time of screening;
* Received lipophilic iodine contrast agents (such as iodized oil, iodized benzene, etc.) within the past 3 months or received water-soluble iodine contrast agents (such as iohexol, iodinated glycerol, etc.) within the past 1 month prior to screening;
* Pregnant or lactating women, or women who engaged in unprotected sexual intercourse within the two weeks prior to screening, or women with a positive blood pregnancy test at screening;
* Male subjects (or their partners) or female subjects who have plans for fertility or donation of sperm or ova during the entire study period and within 6 months after the end of the study, and who are unwilling to adopt contraceptive measures during the study period and within 6 months after the end of the study;
* Researchers believe that the presence of any condition may harm the subjects or prevent them from meeting or fulfilling the study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of hyroid stimulating hormone elevation | For patients in the experimental group: 24 hours after the second time of recombinant human thyroid stimulating hormone injection; For patients in the no intervention group: 4 to 6 weeks after thyroid hormone withdraw
  The proportion of patients with thyroid stimulating hormone>30 mIU/L
Incidence of Treatment-Emergent Adverse Events | Time interval from start to 3 months after completion of the therapy
  This study will utilize the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 4.0 for toxicity and Serious Adverse Event reporting

SECONDARY OUTCOMES:
Overall response rate | 4 month
  Number of patients achieving a complete response (CR) or partial response (PR) by Response Evaluation Criteria (RECIST v1.1 criteria) in Solid Tumors

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China